CLINICAL TRIAL: NCT05056636
Title: Epidemiological Study of Fabry Disease Screening in Chronic Kidney Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Hsing Wu, Director, Division of Nephrology, Department of Internal Medicine, Kaohsiung Chung Gung Memorial Hospital, Chang Gung Memorial Hospital
Other Study IDs: GZ201711687
Record Dates: First submitted 2021-08-31; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Fabry Disease
Keywords: high risk screening; Chronic kidney disease
MeSH Terms: conditions — Fabry Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Plasma α-Gal A activity; Plasma Lyso-GB3; GLA genetic sequencing. — Screening Visit 1:
  1. Male patient will first screened by enzymatic assay (Cutoff: 1.3 μM /hr)
  2. Female patient will first screened by lyso-GB3 (Cutoff: > 5ng/ml)
  Screening Visit 2:
  If both male and female who has deficient enzymatic level (Cutoff: 1.3 μM /hr) or lyso-GB3 level (Cutoff: > 5ng/ml) respectively, those patients will be confirmed whether they have carried Fabry Disease causing mutation by whom GLA genetic sequencing.

SUMMARY:
Fabry disease is a rare X-linked lysosomal storage disorder caused by deficient activity of the enzyme α-Gal A resulting from mutations affecting the GLA gene.

It is characterized by severe multi-systemic involvement that leads to major organ failure and premature death in affected men and in some women. The α-Gal A deficiency results in progressive accumulation of un-degraded glycosphingolipids, predominantly globotriaosylceramide (Gb3), within cell lysosomes throughout the body.

In patients at the second or third decade, progressive proteinuria, decline in glomerular filtration rate (GFR), and tubular damage occur usually, and renal failure develops in the fourth decade. Life-threatening renal, cardiac, and cerebrovascular diseases are added in later decades.

In addition to that, Fabry disease patient will eventually face end-stage renal disease (ESRD) which was the most common cause of death in Fabry patients before the development of dialysis and renal transplantation. Thus it is critical to identify Fabry patient as early as possible, before reaching the stage of ESRD.

Additionally, early intervention of enzyme replacement therapy for Fabry Disease patient which will help the patient to preserve a better renal function and benefit from treatment outcome.

Apart from that today there is only one study published from Turkey for Fabry disease screening in CKD patient where they have screened 1453 and found that the overall prevalence of Fabry disease in CKD patient was found to be 0.2% , 3/1453 (in which 0.4% in 656 male, 0.0% in 783 female). However, there was no information available within the Asia region thereby a very low Fabry disease awareness and diagnostic awareness among nephrologist in Taiwan.

Therefore in the present study the investigators are aiming to investigate the prevalence of Fabry disease in the CKD population (CKD stage 1 ~ 5) by conducting the first and largest high risk screening prevalence study among 2,000 CKD patients over 3 years in Taiwan and the investigators hope by doing such a pilot study our data would contribute to a new paradigm of Fabry disease diagnosis in the Asia region.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 y/o (No age limit due to cardiac variant Fabry IVS4 in Taiwan symptom of onset could be beyond 60 y/o)
* Patient with confirmed chronic kidney disease (CKD 1~5) diagnosis whose urine protein/creatinine (UPCR) is 150mg/g or above, or urine albumin/creatinine (ACR) is 30mg/g or above.
* Patient who are willing to sign inform consent form

Exclusion Criteria:

* Patient who are unwilling to sign inform consent form
* Patient who received confirmed diagnosis of Fabry Disease
* Patient with known etiology of renal failure diagnosed with renal biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2000 Chronic Kidney Disease patient
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive screening rate of Fabry Disease patient among CKD population | 48 months
  Identify the prevalence rate of Fabry disease in patients with CKD including dialysis in Taiwan.

SECONDARY OUTCOMES:
Characterization of gene mutation pattern of Fabry patients with CKD in Taiwan | 48 months
  Identify what gene mutation(s) is(are) significant associated with Fabry patients with CKD in Taiwan

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsing Wu, Principal Investigator — Chang Gung Memory Hospital
Locations (1):
- Chang Gung Memory Hospital, Kaohsiung City, Taiwan